CLINICAL TRIAL: NCT02254499
Title: Prospective Descriptive Study of Nociceptive and Psychological Prediction of Pain After Total Knee Arthroplasty (TKA)
Brief Title: Prediction of Pain After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Iben Engelund Luna, Research Fellow, Rigshospitalet, Denmark
Other Study IDs: H-3-2014-090
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite improvements in treatment, a significant part of patients have severe pain following knee arthroplasty. Preoperative identification of high-risk patients would allow for an intensive individualized analgesic treatment pre- and postoperatively and thus potentially in reduced pain acute and chronically.

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral TKA
* caucasian
* 50 - 80 years
* osteoarthritis

Exclusion Criteria:

* deficient written or spoken danish
* impairment from psychological og neurological disease
* expected discharged to rehabilitation facility
* anticoagulant therapy
* allergies to analgesic treatment
* hypertension (systolic > 160 / diastolic > 100)
* ASA class ≥ 4

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis referred for total knee arthroplasty.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours postoperatively
  Pain intensity on a NRS from 0 to 10 upon ambulation 24 hours following surgery

SECONDARY OUTCOMES:
Pain | 48 hours postoperatively
  Pain intensity on a NRS (numeric rank scale) from 0 to 10 upon ambulation 48 hours following surgery
Pain | From day 1 to day 14 following surgery
  Daily diary reported pain intensity on a NRS (numeric rank scale) from 0 to 10 in average and when worse the first two weeks following knee arthroplasty.

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark